CLINICAL TRIAL: NCT04751331
Title: Neural Response to Inflammatory Challenge in Major Depressive Disorder
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2020-004-00
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LPS (Experimental): Lipopolysaccharide (LPS) (0.8ng/kg of body weight; E. coli group O:113) administered as an intravenous bolus.
  Interventions: Biological: LPS
- Placebo (Placebo Comparator): Placebo (same volume of 0.9% saline) administered as an intravenous bolus
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: LPS — Lipopolysaccharide (LPS) (0.8ng/kg of body weight; E. coli group O:113)
  Arms: LPS
Biological: Saline — 0.9% saline administered as an intravenous bolus
  Arms: Placebo

SUMMARY:
This is a parallel group, double-blinded, placebo-controlled study. Participants with MDD (n=90) and HC (n=90) will be randomly assigned (2:1) to receive either lipopolysaccharide (LPS) (0.8ng/kg of body weight) or placebo (same volume of 0.9% saline) administered as an intravenous bolus. This will yield the following groups: MDD-LPS (n=60), MDD-Placebo (n=30), HC-LPS (n=60), HC-placebo (n=30).

There are three main aims: to identify immune pathways and neural circuits that respond differently to LPS in MDD vs. HC subjects; (2) to test whether the strength of inflammatory changes induced by LPS is associated with degree of change in anhedonic symptoms and neural circuits in the MDD group, and (3) to identify a biotype of MDD that shows a differential immunological and neurophysiological response to LPS. The main outcome variables are symptoms of anhedonia measured with the Snaith-Hamilton Pleasure Scale (SHAPS), cytokines (Il-6, IL-8, IL-10, and TNF), and BOLD signal change in the neural circuitry mediating interoceptive processing, i.e. the insula and cingulate cortex. The exploratory aim is to determine whether the acute inflammatory response to LPS can predict the clinical course of depression over a period of six months. The main outcome of this component of the study is self-reported depressive symptoms assessed with the QIDS-SR.

DETAILED DESCRIPTION:
This is a parallel group, double-blinded, placebo-controlled study. Participants with MDD (n=90) and HC (n=90) will be randomly assigned (2:1) to receive either lipopolysaccharide (LPS) (0.8ng/kg of body weight; E. coli group O:113) or placebo (same volume of 0.9% saline) administered as an intravenous bolus. This will yield the following groups: MDD-LPS (n=60), MDD-Placebo (n=30), HC-LPS (n=60), HC-placebo (n=30). Individuals who are eligible for the study will be randomly assigned through the use of a block randomization scheme to ensure the inclusion of equal numbers of HC and MDD participants in each group. MDD participants will complete up to 10 study visits (V1-V10) while the HCs will complete up to four visits (V1-V4). At visit 1 (V1), each subject will be consented and will complete the following: self-report and clinician-administered scales (including the Columbia Suicide Severity Rating Scale), a physical exam that includes an EKG and vital signs (temperature, pulse, blood pressure), safety labs (CBC, CMP, TSH, HbA1C, HIV, HCV), a urine drug screen, an alcohol breathalyzer, and a baselineMRI session comprising the following scans: clinical, anatomical, visceral interoceptive attention (VIA) task, monetary incentive delay task (MID) and resting state fMRI. Vital signs will be assessed in a supine position with a completely automated device. Blood pressure and heart-rate measurements will be preceded by at least five minutes of rest in a quiet setting without distractions. Blood will be drawn via venipuncture using sterile techniques by a trained phlebotomist or nurse.

Subjects that pass the safety screen return two days later for the experimental session (V2). Prior to infusion of LPS or saline, the Columbia, EKG, urine drug screen, and breathalyzer are repeated, vital signs are taken, and baseline (T0) rating scales and blood draws are completed. A nurse will insert a catheter with a heparin lock into the non-dominant forearm for blood draws and a continuous saline flush, and one into the dominant forearm for LPS or saline administration. Prior to the LPS/saline infusion, participants will be hydrated with 500cc of saline. The LPS to be used in the study will be obtained from the NIH Clinical Center. Vital signs will be assessed every 30 min post infusion of LPS/saline for the first 2 hours (and thereafter every hour). Blood samples will be taken at baseline (T0), at T1 and then at T1.5 and T3.5 (~ peak response) and prior to discharge at T6. Participants also will complete hourly measures of sickness symptoms (e.g., fatigue, pain), anxiety, depression, and anhedonia. Symptoms will be recorded and graded according to FDA criteria. Two hours post-infusion at the approximate peak of the inflammatory response, the participants will complete the same MRI scans as at baseline. Subject to the judgment of a physician, the participants will be discharged 6 hours post injection so that the total experimental procedure will take ~8 hours to complete. Participants return the following day (T24) and one week later (V4) for mood ratings, blood draws, and identical MRI sessions. MDD participants will also be followed longitudinally for 6 months (phase 2), in the process completing remote or in-person psychological assessments at months 1 through 6 post LPS-infusion.

Participants will be recruited from the Tulsa metropolitan area through internet, radio, print advertisements and will be evaluated at LIBR. We may also advertise the study to students on Tulsa-area campuses using flyers and potentially also recruitment tables on campus, and discussions with organizations, classes, and faculty where permission from the appropriate university officials is obtained. A total of 200 human participants (180 completers of phase I) will be involved in the proposed research. Half the participants will be males or females between the ages of 18 and 65 with MDD and current symptoms of depression (mild to severe) and half the participants will be HC with no personal history of psychiatric illness. A DSM-V diagnosis of MDD will be made with the MINI International Neuropsychiatric Interview and current symptoms of depression will be measured with the clinician-administered Montgomery Asberg Depression Rating Scale (MADRS), the self-report Patient Health Questionnaire (PHQ-9), and the Quick Inventory of Depressive Symptoms (QIDS-SR). Depressed participants will be required to be in good general health (as evaluated during the screening visit, including physical exam, safety labs and EKG) and to be 18-65 years of age. MDD participants will be required to have symptoms of depression, that is, a MADRS score of ≥7 or a PHQ-9 score ≥10. MDD participants are also required to be unmedicated for at least 4 weeks (8 weeks for fluoxetine) or currently receiving treatment with only one anti-depressant medication. HC participants will be required to be in good general health and to be 18-65 years of age.

There are three main aims: to identify immune pathways and neural circuits that respond differently to LPS in MDD vs. HC subjects; (2) to test whether the strength of inflammatory changes induced by LPS is associated with degree of change in anhedonic symptoms and neural circuits in the MDD group, and (3) to identify a biotype of MDD that shows a differential immunological and neurophysiological response to LPS. The main outcome variables are symptoms of anhedonia measured with the Snaith-Hamilton Pleasure Scale (SHAPS), cytokines (Il-6, IL-8, IL-10, and TNF), and BOLD signal change in the neural circuitry mediating interoceptive processing (the insula and cingulate cortex), and BOLD signal change in the neural circuitry mediating reward (ventral striatum). The exploratory aim is to determine whether the acute inflammatory response to LPS can predict the clinical course of depression over a period of six months. The main outcome of this component of the study is self-reported depressive symptoms assessed with the QIDS-SR.

ELIGIBILITY:
Inclusion Criteria:

Both healthy controls and depressed participants will be required to be in good general health (as evaluated during Visit 1, including EKG) and to be 18-65 years of age. A DSM-V diagnosis of MDD will be made with the MINI International Neuropsychiatric Interview and current symptoms of depression will be measured with the clinician-administered MADRS and the self-report PHQ-9. Depressed participants will be required to have symptoms of depression (i.e. a PHQ-9 score ≥10) and/or a MADRS score of ≥7.

Exclusion Criteria:

General Exclusion Criteria:

* Pregnancy
* A history of fainting during blood draws will be evaluated by the clinical team and may be deemed exclusionary.

Medical Conditions:

* Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits.
* Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders.
* Presence of co-morbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders.
* Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk.
* Presence of chronic infection that may elevate pro-inflammatory cytokines.
* Presence of an acute infectious illness or receipt of a vaccination in the two weeks prior to an experimental session.

Psychiatric Disorders:

* Current severe suicidal ideation or attempt within the past 12 months.
* Psychosis
* Bipolar disorder
* Substance abuse or dependence within the previous 6 months

Contraindications for MRI:

* Cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.
* Claustrophobia that is severe enough to preclude MRI scanning.

Medications:

* Current and/or past regular use of hormone-containing medications (excluding contraceptives)
* Use of medications such as oral corticosteroids which may have immunosuppressive effects.
* Current use of non-steroid anti-inflammatory drugs that is deemed by the investigators to potentially confound the results of the study (e.g. > 3 days/week)
* Current and/or past regular use of immune modifying drugs that target specific immune responses such as TNF antagonists
* Current use of analgesics such as opioids or history of addiction to opioids or other analgesics
* Current and/or past regular use of cardiovascular medications, including antihypertensive, antiarrhythmic, anti-anginal, and anticoagulant drugs (does not apply where medications are taken for different purpose e.g. anti-hypertensives for migraine).
* Chronic use of antibiotics such as isotretinoin or minocycline because of their potential effects on the microbiome and immune function.
* Evidence of recreational drug use from urine test.
* Lifetime use of methamphetamine
* Inclusion of individuals reporting other types of medications or supplements not listed or considered thus far will be at the discretion of the PI based on their potential to affect immune function, the microbiome, brain function or brain blood flow.

Health Factors:

* BMI > 35 because of the effects of obesity on pro-inflammatory cytokine activity
* Clinically significant abnormalities on screening laboratory tests
* Abnormal EKG
* In addition, participants who on arrival to the study, show any of the following symptoms will not be allowed to complete the study:

  1. screening supine systolic blood pressure >140 mmHg or <100 mmHg
  2. screening supine diastolic blood pressure >90 mmHg or <60 mmHg
  3. 12-lead EKG demonstrating a PR interval > 0.2 msec QTc >450 or QRS >120 msec (Bazett) If the QTc exceeds 450 msec, or QRS exceeds 120 msec, the EKG will be repeated 2 more times and the median value will be used
  4. pulse less than 50 beats/minute or greater than 100 beats/minute
  5. temperature greater than 99.5 degrees F.

     Non-English speaking participants:
* The majority of the assessments proposed for this study have not been translated from English, thus, non-English speaking volunteers will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Inflammatory response | 1.5 hours post infusion
  Serum interleukin 6 (IL-6) (pg/mL)

SECONDARY OUTCOMES:
Symptoms of anhedonia | 1.5 hours post infusion
  Snaith-Hamilton Pleasure Scale Score (score range 14-56; higher scores more anhedonia)
Depressive Symptoms | 24 hours post infusion
  Change in Depressive Symptoms measures with the Montgomery-Asberg Depression Rating Scale (MADRS). Score range 0-60. Higher scores = more depression.
Neural response to anticipation of monetary reward | Two hours post-infusion
  BOLD Signal Change in the ventral striatum measured using MRI
Neural response to interoceptive vs exteroceptive stimuli (interoceptive awareness task) | Two hours post infusion
  BOLD Signal Change in the Insula and Posterior Cingulate Cortex measured using MRI

OTHER OUTCOMES:
Temperature | 3-5 hours post infusion
  Body temperature
Inflammatory response | 1.5 hours post-infusion
  Serum tumor necrosis factor (TNF) (pg/mL)
Course of Illness | 6 months
  Depressive symptoms at 6 month follow-up measured with the Quick Inventory of Depressive Symptoms (QIDS). Score range 0-27. Higher scores = greater depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04751331/ICF_001.pdf